CLINICAL TRIAL: NCT03144297
Title: Correlation Between Intracranial Pressure as Measured by Lumbar Puncture Manometry and Percentage Body Fat as Measured by Air-displacement Plethysmography
Brief Title: Intracranial Pressure vs Percentage Body Fat
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Benjamin Wakerley, Consultant neurologist, Gloucestershire Hospitals NHS Foundation Trust
Other Study IDs: 14/LO/2266
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Intracranial Pressure
MeSH Terms: interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lumbar puncture — diagnostic lumbar puncture
Other: BOD POD (air-displacement plethysmography) — Assessment of body fat

SUMMARY:
Background: It has already been established that there is a weak positive relationship between increased intracranial pressure (ICP), as measured by lumbar puncture manometry, and increased Body Mass Index (BMI). This is also observed clinically in some patients with idiopathic intracranial hypertension, who typically have raised BMI. The relationship between BMI and percentage body fat is non-linear, especially at BMI > 40. The Bod Pod device enables non-invasive body composition profiling, including accurate calculation of percentage body fat, without the use of radiation.

Aim: To examine the relationship between intracranial pressure as measured by lumbar puncture manometry and percentage body fat as measured by air-displacement plethysmography (Bod Pod)

Methods: 100 patients undergoing routine diagnostic and therapeutic lumbar punctures for a variety of non-emergency neurological conditions will be recruited. Cerebrospinal fluid opening pressure will be measured using standard manometry techniques. Blood pressure, height, weight, collar size, waist size and hip size will be measured. Body composition profiling will be carried out using the Bod Pod.

DETAILED DESCRIPTION:
Patients due to attend the elective lumbar puncture clinic will be contacted by letter beforehand (at least a week) and provided with an information sheet about the this study. Neurology patients are referred to the lumbar puncture clinic as part of their diagnostic work-up. The clinic takes place every Friday on the neurology ward and is run by the MS nurse consultant who does the procedure.

Patients agreeing to take part in the study will have a lumbar puncture as normal. Before removing a small volume of spinal fluid (cerebrospinal fluid or CSF), the investigators routinely measure spinal fluid pressure using a manometer (pressure gauge). This is important because it indirectly tells us what the pressure is within the brain (intracranial pressure or ICP). Samples of CSF and blood may be needed as part of NHS patient care, but no additional samples will be needed for this study. The investigators will, however, take some additional measurements during the visit, which won't take more than an extra 5 minutes. These will include: weight and height; measures of neck, waist and hip circumference, using a standard measuring tape; and blood pressure before and after the lumbar puncture. The whole visit will be 45-60 minutes.

Patients agreeing to have body composition assessment in the Bod Pod device will be scheduled for assessment at the School of Sport Sciences at the University of Gloucestershire (Oxstalls campus) in the two weeks following lumbar puncture. The investigators will also contact patients prior to the appointment to confirm this. The university is a five minute drive from the hospital and can easily be accessed by public transport. Temporary parking permits for use in the university car park will be provided where necessary. At the university body composition will be assessed in the Bod Pod device by one of the trained technicians. The device consists of a small enclosed chamber, in which the patient sits. Changes in air volume allow calculation of body density and percentage body fat. For the test, patients will need to bring some form of tight-fitting swimwear (Speedos or underpants for men; swimming costumes for women, no bikinis). They will also be required to wear a swimming hat (which will be provided). No metal objects should be worn while in the Bod Pod. Prior to the test we may need to measure lung volume by asking the patient to blow into a spirometer. This helps to calculate body density but is not always necessary. The patient will then sit inside the Bod Pod (which is confined but non-invasive and has a large window in the front hatch and a panic button if they want to alert the technician) for about 3 minutes. During this time air displacement measurements are made and some people may experience slight pressure in their ears, although this is not dangerous. Male and female changing facilities are available and Bod Pod testing will be in a private, screened-off area with only the technician present. Patients can also ask for a chaperone or male/female technician if they prefer. This test will take about 15 minutes to complete and patients will be given computer readout of their body composition.

A power calculation for the study indicates that approximately 100 patients will need to be recruited. The investigators aim to recruit between 1 and 3 patients from the lumbar puncture clinic per week and therefore predict that the study will be completed within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects recruited from general neurology clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Intracranial pressure vs % body fat using BodPOD | 3 years
  Correlation between intracranial pressure as measured by lumbar puncture manometry and percentage body fat as measured by air-displacement plethysmography.

SECONDARY OUTCOMES:
intracranial pressure vs body mass index | 3 years
  Correlation between intracranial pressure as measured by lumbar puncture manometry and body mass index.

CONTACTS AND LOCATIONS:
Locations (1):
- Benjamin Wakerley, Gloucester, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No